CLINICAL TRIAL: NCT02259699
Title: Ovarian Cancer Patient-Centered Decision Aid
Acronym: PCOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Lari Wenzel, Professor of Medicine, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PCORI CE-12-11-4755
Record Dates: First submitted 2014-05-15; First posted 2014-10-08 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Stage III Ovarian Cancer
Keywords: Ovarian Cancer; Intraperitoneal chemotherapy; Intravenous chemotherapy; decision making
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Aid (PCOA) (Experimental): PCOA will be designed to accomplish 2 objectives: 1) it will educate patients and allow them to assimilate information about the differences in outcomes and survival between IP and IV therapies; and 2) it will help patients make the difficult trade-offs between these two treatment options.
  Interventions: Other: Decision Aid
- UC (Standard care) (No Intervention): Standard pamphlets will be given to patients to educate them about IV and IV/IP therapies.

INTERVENTIONS:
Other: Decision Aid — PCOA will be designed to accomplish 2 objectives: 1) it will educate patients and allow them to assimilate information about the differences in outcomes and survival between IP and IV therapies; and 2) it will help patients make the difficult trade-offs between these two treatment options.
  Other Names: Patient Centered Outcome Aid (PCOA)
  Arms: Decision Aid (PCOA)

SUMMARY:
The objective of this study is to develop and test a new decision aid -named Patient Centered Outcome Aid (PCOA)-that will allow patients to assimilate information and identify trade-offs about the impact of IP/IV therapy versus IV-only therapy on their QOL and survival, based on their own preferences and personal clinical characteristics, described in terms that are meaningful to them. To accomplish this, the investigators will 1)develop the PCOA, a patient- and provider-friendly decision aid and 2)test the effectiveness of PCOA through a randomized controlled trial (RCT).

The investigators hypothesize that PCOA will be significantly better than usual care, resulting in patients reporting more satisfaction with their treatment decision, less decision regret, better quality of life, and more satisfaction with their care compared with similar patients not having access to PCOA. If these hypotheses are substantiated, patients and providers will have an improved model for communication and decision making, leading to better patient outcomes.

DETAILED DESCRIPTION:
Ovarian cancer is typically diagnosed at an advanced stage and carries the highest fatality-to-case ratio of all gynecologic malignancies diagnosed in the United States. Arguably the most effective treatment regimen to date is provided through intraperitoneal (IP) chemotherapy delivery, together with intravenous (IV) chemotherapy, which in the most recent phase III randomized trial conferred the longest median survival (65.6 months) ever reported in advanced ovarian cancer, compared to 49.7 months in the IV-only treatment arm. However, during active treatment, patients randomized to the IP therapy group reported significantly worse quality of life (QOL), and more treatment-related toxicities. In short, women are less likely to die if they receive an IP component to their chemotherapy, a finding that was underscored by an NCI Clinical Alert. However, there may be greater toxicity with IP treatment. The tradeoff between short-term reduced QOL and longer survival is difficult for patients to understand and then incorporate meaningfully into their decision-making process. In fact, for reasons that are not entirely clear, many patients are not offered IP therapy. Patient-centered care requires that they be given the opportunity to participate in treatment decision-making.

ELIGIBILITY:
Inclusion Criteria:

* RCT participants will include stage III optimally debulked advanced ovarian cancer patients from urban and rural regions of the country, who will be randomized to either our patient-centered decision-aid or the usual care control arm

Exclusion Criteria:

* By the nature of the neoplasm under study, gender specific (ovarian cancer), only female patients will be included
* Patient enrollment will include women from all English speaking ethnic groups

  -> the age of 21
* All minority ovarian cancer survivors will be eligible
* Women under age 21 will not be included in this study because it is not common to be diagnosed with advanced epithelial ovarian cancer in females under age 21

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lari Wenzel, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Decision Aid (PCOA) | UC (Standard Care)
Started | 64 | 60
Completed | 37 | 40
Not Completed | 27 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid (PCOA) | UC (Standard Care) | Total
Number analyzed (Participants) | 64 | 60 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 45 | 89
  >=65 years | 20 | 15 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (11.0) | 58.2 (8.8) | 58.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 60 | 124
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 64 | 60 | 124

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Decision
Description: Satisfaction with Decision scale (SWD) is a 6-item scale measuring satisfaction with health care decisions, developed and validated in the context of women making decisions about hormone replacement therapy, and subsequently validated in adults with depression making decisions about treatment. The scale has good internal consistency reliability (alpha = 0.85), evidence of construct validity, relevance to designing and assessing patient-centered decision support interventions, and is sensitive to changes in information in trials of decision aids. The scale uses a 1-5 rating (1=strongly disagree; 5 = strongly agree). Scores from these 6 items were linearly transformed to a 0-100 scale. A higher score reflects a higher level of satisfaction with the decision.
Time Frame: at treatment initiation (T1), treatment completion (T3), and 9 months post enrollment (T4)
Population: Includes 63 PCOA and 56 UC with complete data
Measure: Mean (Standard Error); unit: transformed scale score
Arm/Group | Decision Aid (PCOA) | UC (Standard Care)
Number analyzed (Participants) | 63 | 56
transformed scale score
  T1 | 85.3 (2.0) | 86.9 (2.1)
  T3: number analyzed (Participants) | 49 | 52
  T3 | 85.8 (2.1) | 91.5 (2.0)
  T4: number analyzed (Participants) | 37 | 40
  T4 | 87.1 (2.4) | 90.6 (2.3)
Statistical Analysis 1: Comparison: Decision Aid (PCOA) vs UC (Standard Care); Difference between arms at T1; Test type: Superiority; p = 0.582, t-test, 2 sided
Statistical Analysis 2: Comparison: Decision Aid (PCOA) vs UC (Standard Care); Difference between arms at T3; Test type: Superiority; p = 0.053, t-test, 2 sided
Statistical Analysis 3: Comparison: Decision Aid (PCOA) vs UC (Standard Care); Difference between arms at T4; Test type: Superiority; p = 0.288, t-test, 2 sided

2. Primary Outcome: Decisional Regret
Description: The Decision Regret Scale is a 5-item scale which is a reliable and valid indicator of health care decision regret at a given point in time, with excellent psychometric properties. In this study, the question stem will ask "about the decision you made about selecting IP/IV treatment." Total scores were linearly transformed to a 0-100 scale. The lowest possible score, 0, means no regret. The highest possible score, 100, means high regret. This outcome will be measured from T2 - T4, but is not appropriate to ask at the time of the T1 assessment, which is just after the treatment decision has been made, but prior to treatment delivery. Use of this measure will allow us to evaluate whether the PCOA, compared to usual care, helps to reduce regret during and after cancer treatment.
Time Frame: At treatment completion (T3) and 9 months post enrollment (T4)
Population: Includes 48 PCOA and 52 UC with complete data at T3
Measure: Mean (Standard Error); unit: transformed scale score
Arm/Group | Decision Aid (PCOA) | UC (Standard Care)
Number analyzed (Participants) | 48 | 52
transformed scale score
  T3 | 16.6 (2.0) | 11.7 (1.9)
  T4 | 15.4 (2.6) | 15.0 (2.5)
Statistical Analysis 1: Comparison: Decision Aid (PCOA) vs UC (Standard Care); Difference between arms at T3; Test type: Superiority; p = 0.087, t-test, 2 sided
Statistical Analysis 2: Comparison: Decision Aid (PCOA) vs UC (Standard Care); Difference between arms at T4; Test type: Superiority; p = 0.910, t-test, 2 sided

3. Secondary Outcome: Shared Decision Making
Description: The 9-item Shared Decision Making Questionnaire (SDM-Q-9) was developed and psychometrically tested for use in clinical encounters. It has strong reliability and validity, and use is advocated in studies investigating the effectiveness of interventions aimed at implementing shared decision-making. The question stem indicated the medical decision (IP/IV) with 6 levels of agreement from 'completely disagree to completely agree' (e.g., "My doctor and I selected a treatment option together"). Total scores were linearly transformed to range from 0 to 100, where 0 indicates the lowest possible level of SDM and 100 indicates the highest extent of SDM. SDM was assessed at T1 only, since this was the most proximal in time to when the decision was made.
Time Frame: at treatment initiation (T1)
Population: Includes 63 PCOA and 56 UC with complete data
Measure: Mean (Standard Error); unit: tansformed scale score
Arm/Group | Decision Aid (PCOA) | UC (Standard Care)
Number analyzed (Participants) | 63 | 56
tansformed scale score | 79.5 (2.2) | 78.7 (2.6)
Statistical Analysis 1: Comparison: Decision Aid (PCOA) vs UC (Standard Care); Test type: Superiority; p = 0.807, t-test, 2 sided

4. Secondary Outcome: Satisfaction With Care (EORTC) Overall Quality Rating
Description: Satisfaction with Care was measured using the EORTC IN-PATSAT32, which assessed cancer patients' appraisal of doctors and nurses, as well as aspects of care organization and services. The measure also discriminated between cancer patients with different care expectations. Scores from these 32 items were linearly transformed to a 0-100 scale. A higher score reflects a higher level of satisfaction. This measure has excellent internal consistency and convergent validity, although some scales are highly correlated. Test-retest reliability is acceptable.
Time Frame: at treatment completion (T3) and 9 months post enrollment (T4)
Population: Includes 48 PCOA and 52 UC with complete data at T3
Measure: Mean (Standard Error); unit: tansformed scale score
Arm/Group | Decision Aid (PCOA) | UC (Standard Care)
Number analyzed (Participants) | 48 | 52
tansformed scale score
  T3 | 84.4 (3.0) | 90.9 (1.9)
  T4: number analyzed (Participants) | 37 | 40
  T4 | 82.4 (3.5) | 86.9 (3.0)
Statistical Analysis 1: Comparison: Decision Aid (PCOA) vs UC (Standard Care); Difference between arms at T3; Test type: Superiority; p = 0.071, t-test, 2 sided
Statistical Analysis 2: Comparison: Decision Aid (PCOA) vs UC (Standard Care); Difference between arms at T4; Test type: Superiority; p = 0.332, t-test, 2 sided

5. Secondary Outcome: Cancer Therapy Satisfaction
Description: While the EORTC IN-PATSAT32, assessed cancer patients' appraisal of doctors, nurses, and services, the Satisfaction with Cancer Treatment Questionnaire assessed patients' satisfaction specifically with their most recent therapy (i.e. IV or pills). The scale contained 21 items assessing seven domains. Total scores were linearly transformed to a 0-100 scale. A higher score reflects a higher level of satisfaction with their most recent therapy.
  This has been validated on adults with many cancer types and treatments.
Time Frame: at treatment completion (T3) and 9 months post enrollment (T4)
Population: Includes 48 PCOA and 52 UC with complete data at T3
Measure: Mean (Standard Error); unit: tansformed scale score
Arm/Group | Decision Aid (PCOA) | UC (Standard Care)
Number analyzed (Participants) | 48 | 52
tansformed scale score
  T3 | 81.9 (1.9) | 85.8 (2.1)
  T4: number analyzed (Participants) | 37 | 40
  T4 | 83.0 (2.4) | 81.9 (3.0)
Statistical Analysis 1: Comparison: Decision Aid (PCOA) vs UC (Standard Care); Difference between arms at T3; Test type: Superiority; p = 0.177, t-test, 2 sided
Statistical Analysis 2: Comparison: Decision Aid (PCOA) vs UC (Standard Care); Difference between arms at T4; Test type: Superiority; p = 0.745, t-test, 2 sided

6. Other Pre Specified Outcome: Process Outcome - Satisfaction With PCOA Aid
Description: Usability and acceptability of PCOA data will be gathered only from the intervention arm. The usability and acceptability of the PCOA program will be determined both through objective data gathered as patients use the application, and through subjective data gathered through a short, self-report survey that will appear on the PCOA application at the end of the session.
Time Frame: at treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid (PCOA)
Number analyzed (Participants) | 52
Participants
  Very satisfied | 17
  Quite a bit satisfied | 19
  Somewhat satisfied | 15
  A little bit satisfied | 1
  Not at all satisfied | 0

ADVERSE EVENTS:
Description: Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Decision Aid (PCOA) | UC (Standard Care)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No